CLINICAL TRIAL: NCT06283173
Title: Human Repeat Insult Patch Test (HRIPT): Assessment of Primary and Cumulative Skin Irritation and Skin Sensitization of a Product, Under Controlled and Maximized Conditions
Brief Title: HRIPT for Collagen Dressing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Covalon Technologies Inc. (Industry)
Collaborators: ALS Beauty and Personal Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-401
Record Dates: First submitted 2024-02-22; First posted 2024-02-28 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Skin Sensitisation

STUDY DESIGN:
Intervention Model Description: This will be a single center, with no randomization or blinding, study design in 50 healthy adult subjects, age 18-70 years. Based on prior experience approximately 75 subjects will be enrolled to ensure 50 subjects complete the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Collagen wound dressing with positive and negative controls (Experimental): Application of test dressing, 0.5% sodium lauryl sulfate in distilled water, and distilled water on areas of the back or upper arm.
  Interventions: Device: ColActive Plus Collagen Matrix Dressing

INTERVENTIONS:
Device: ColActive Plus Collagen Matrix Dressing — Induction phase: Test article applied with Hill Top chamber every 48+ hours over 3 weeks. Rest phase: 10-day rest period with no application.
  Challenge phase: Test article applied for 48 hours and evaluated through 48 hours post removal.
  The positive control is evaluated at Induction 1 only. The negative control is applied following the same schedule as the test article.

SUMMARY:
The objectives of this study are to determine by repetitive epidermal contact, the primary or cumulative irritation and the allergic contact sensitization potential of the ColActive Plus Collagen Matrix Dressing, under maximized conditions, with controlled product quantity and application site.

DETAILED DESCRIPTION:
Approximately 75 healthy subjects satisfying all criteria listed below will be enrolled to complete the study with a minimum of 50 subjects. The test product will be applied on the 25-millimeter Hill Top Chamber®, which will be applied directly to the test site. The positive control will be applied to each subject for the first 48 hours only, and the negative control will be applied throughout the study along with the test product. Enough product will be used to cover the chamber. The procedure involves occlusive patching of the test product and control(s) for a minimum of 48 hours followed by an assessment. The procedure will be repeated until a series of 9 consecutive 48-hour exposures have been made over 3 consecutive weeks. This induction phase is followed by an approximate two-week rest period. The challenge phase consists of a challenge or test dose applied once to a previously unexposed test site. Clinical staff will remove the patches 48 hours post-application. Reactions will be scored 30 minutes post-removal, 24-hours post-removal, and 48-hours post-removal. Skin response at each application site will be evaluated according to the Berger and Bowman Scale.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70
2. Sex: Male & Female
3. Fitzpatrick: I-V, minimum 10% of panel Fitzpatrick V.
4. Individuals who will be able to read, understand and give an informed consent relating to the study they are participating in.
5. Individuals who will be free of any dermatological or systemic disorder, which in the Investigator's opinion, could interfere with the study results.
6. Individuals who will be in general good health and who will complete a preliminary medical history form mandated by the testing facility.
7. Individuals who will be able to and agree to cooperate with the Investigator and clinical staff.
8. Individuals who will agree to have test products applied in accordance with the protocol and are able to complete the full course of the study.
9. Individuals who have not participated in a similar study in the past 30 days.
10. Individuals who agree to refrain from sun tanning/bathing and prolonged exposure to sunlight (outdoors).
11. Female volunteers who are willing to undergo a urine pregnancy test.
12. Individuals who agree to not change their current brand of personal care products such as soaps, body washes, laundry detergents, body sprays, body spritzes, etc. while participating on the study.

Exclusion Criteria:

1. Individuals who are currently taking any medications (topical or systemic) that may mask or interfere with the test results (specifically, corticosteroids, topical and/or systemic [except nasal steroids], non steroidal anti-inflammatory drugs [e.g. ibuprofen, Advil, Motrin, aspirin > 325mg/day], antihistamines, and topical/oral immunosuppressive medications). Subjects must refrain from using any topical/oral anti-inflammatory medications during the length of the study (6 weeks).
2. Individuals who have a history of any acute or chronic disease that might interfere with or increase the risk on study participation. (e.g., systemic lupus erythematosus, rheumatoid arthritis, HIV positive).
3. Individuals who are diagnosed with chronic skin allergies (atopic dermatitis/eczema) or recently treated skin cancer within the last 12 months.
4. Individuals who have damaged skin in close proximity to test sites (e.g., sunburn, uneven skin pigmentation, tattoos, scars, excessive hair, active acne papules or other disfigurations).
5. Individuals who control their diabetes using insulin.
6. Individuals with any history, which in the Investigator's opinion, indicates the potential for harm to the subject or places the validity of the study in jeopardy.
7. Female volunteers who indicate that they are pregnant or are planning to become pregnant or nursing.
8. Individuals with a known history of hypersensitivity to any cosmetics, personal care products, fragrances, and/or adhesives.
9. Employees of ALS.
10. Individuals with a known fish allergy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan DeSantis, MHI, BS, Principal Investigator — ALS
Locations (1):
- ALS Beauty and Personal Care, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bowman JP, Berger RS, Mills OH, Kligman AM, Stoudemayer T. The 21-day human cumulative irritation test can be reduced to 14 days without loss of sensitivity. J Cosmet Sci. 2003 Sep-Oct;54(5):443-9. PMID 14605686

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects receive the positive control, negative control and test product at the same time. The positive control is only applied at the first visit to ensure the subject responds appropriately to a sensitizer. From then on, both the negative control and test products are applied at the same times at different sites, and both sites are evaluated for a local reaction.
Groups:
- Test Article (Collagen Wound Dressing) and Negative Control (Distilled Water): Each subject will be treated with an occlusive patch of the test article (collagen dressing) and the negative control (distilled water) at the same time.
  During the induction phase of the study, the test article and negative control will be applied repetitively and continuously on one side of the paraspinal region of the back. Each application will be for approximately 48 hours (weekdays) or 72 hours (weekends) over three weeks for a total of 9 applications. During a subsequent challenge phase at least 10 days after the induction phase, the test article and negative control will be applied for 48 hours. The application sites of the subject will be evaluated at approximately 30 minutes, 24 hours, and 48 hours after removal of the test article and negative control.
Period: Overall Study
Arm/Group | Test Article (Collagen Wound Dressing) and Negative Control (Distilled Water)
Started | 86
Completed | 57
Not Completed | 29
Not completed — Did not show for first visit | 10
Not completed — Lost to Follow-up | 12
Not completed — Physician Decision | 7

BASELINE CHARACTERISTICS:
Groups:
- Collagen Wound Dressing With Positive and Negative Controls: Application of test dressing, 0.5% sodium lauryl sulfate in distilled water, and distilled water on areas of the back or upper arm.
  ColActive Plus Collagen Matrix Dressing: Induction phase: Test article applied with Hill Top chamber every 48+ hours over 3 weeks. Rest phase: 10-day rest period with no application.
  Challenge phase: Test article applied for 48 hours and evaluated through 48 hours post removal.
  The positive control is evaluated at Induction 1 only. The negative control is applied following the same schedule as the test article.
Arm/Group | Collagen Wound Dressing With Positive and Negative Controls
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African American | 18
  Race: Asian | 10
  Race: Caucasian | 11
  Race: Hispanic | 14
  Race: Other | 4
Region of Enrollment [Number; unit: participants]
  United States | 57
Fitzpatrick Skin Type [Count of Participants; unit: Participants]
  I - always burn, does not tan | 3
  II - burn easily, tan slightly | 14
  III - burn moderately, tan progressively | 10
  IV - burn a little, always tan | 13
  V - rarely burn, tan intensely | 17
  VI - never burn, tan very intensely | 0

OUTCOME MEASURES:

1. Primary Outcome: Skin Sensitization Reaction Using Berger and Bowman Scale
Description: Inflammatory response graded as 0 through 3: 0=no visible reaction; +=slight, confluent, or patchy erythema; 1=Mild erythema (pink); 2=moderate erythema (definite redness); 3=strong erythema (very intense redness)
  Definition of letter grades appended to a numerical grade:
  E = Edema - swelling, spongy feeling when palpated P = Papule - red, solid, pinpoint elevation V = Vesicle - small elevation containing fluid B = Bulla reaction - fluid-filled lesion (blister) S = Spreading - evidence of the reaction beyond the Webril® pad area W = Weeping - result of a vesicular or bulla reaction - serous exudate I = Induration - solid, elevated, hardened, thickened skin Superficial Effects g = Glazing y = Peeling c = Scab, dried film of serous exudate of vesicular or bulla reaction d = Hyperpigmentation (reddish-brown discoloration of test site) h = Hypopigmentation (loss of visible pigmentation at test site) f = Fissuring - grooves in the superficial layers of the skin
Time Frame: 48 hours post challenge and 24 hours and 48 hours post-challenge removal
Measure: Mean (Full Range); unit: score on a scale
Units Other Than Participants: Skin sites
Groups:
- Test Article (Collagen Wound Dressing): Application of test dressing to test site using a 25-mm Hill Top Chamber. One test dressing will be applied directly to the test site (intrascapular region or upper arm) of the subject at each planned exposure.
- Negative Control (Distilled Water): Application of distilled water to test site using a 25-mm Hill Top Chamber. One negative control will be applied directly to the same test site (intrascapular region or upper arm) of the subject throughout the study following the same protocol as the test product.
Arm/Group | Test Article (Collagen Wound Dressing) | Negative Control (Distilled Water)
Number analyzed (Participants) | 57 | 57
Number analyzed (Skin sites) | 57 | 57
score on a scale
  Mean score at 48 hours post challenge | 0 [0 to 0] | 0 [0 to 0]
  Mean score at 24 hours post challenge removal | 0 [0 to 0] | 0 [0 to 0]
  Mean score at 48 hours post-challenge removal | 0 [0 to 0] | 0 [0 to 0]

2. Other Pre Specified Outcome: Induction Phase Skin Response
Description: Assessment of irritation based on the Berger and Bowman scale:
  Numeric Scores 0 = No evidence of irritation
  1. = Minimal erythema, barely perceptible
  2. = Moderate erythema, readily visible; or minimal edema; or minimal papular response
  3. = Strong erythema; or erythema and papules
  4. = Definite edema
  5. = Erythema, edema and papules
  6. = Vesicular eruption
  7. = Strong reaction spreading beyond test site Letter Grades (always upper case) A = Slight glazed appearance B = Marked glazing C = Glazing with peeling and cracking F = Glazing with fissures G = Film of dried serous exudate covering all or a portion of the patch site H = Small petechial erosions and/or scabs Positive control should show a response and negative control should not show a response.
Time Frame: Every 48-72 hours for 1 (positive control) or 9 (negative control and test) applications
Population: Assessment of the positive control was only planned post-application #1 but was also performed post-application #2.
Measure: Mean (Full Range); unit: score on a scale
Units Other Than Participants: Skin sites
Groups:
- Positive Control (0.5% Sodium Lauryl Sulfate): Application of 0.5% sodium lauryl sulfate to test site using a 25-mm Hill Top Chamber.
  One positive control will be applied directly to a test site (intrascapular region or upper arm) of the subject and will only be applied for Induction 1 (the first 48 hours).
Arm/Group | Test Article (Collagen Wound Dressing) | Negative Control (Distilled Water) | Positive Control (0.5% Sodium Lauryl Sulfate)
Number analyzed (Participants) | 57 | 57 | 57
Number analyzed (Skin sites) | 57 | 57 | 57
score on a scale
  Post-application 1 | 0 [0 to 0] | 0 [0 to 0] | 0.6 [0 to 3]
  Post-application 2 | 0 [0 to 0] | 0 [0 to 0] | 0.5 [0 to 2]
  Post-application 3: number analyzed (Participants) | 57 | 57 | 0
  Post-application 3: number analyzed (Skin sites) | 57 | 57 | 0
  Post-application 3 | 0 [0 to 0] | 0 [0 to 0] |
  Post-application 4: number analyzed (Participants) | 57 | 57 | 0
  Post-application 4: number analyzed (Skin sites) | 57 | 57 | 0
  Post-application 4 | 0 [0 to 0] | 0 [0 to 0] |
  Post-application 5: number analyzed (Participants) | 57 | 57 | 0
  Post-application 5: number analyzed (Skin sites) | 57 | 57 | 0
  Post-application 5 | 0 [0 to 0] | 0 [0 to 0] |
  Post-application 6: number analyzed (Participants) | 57 | 57 | 0
  Post-application 6: number analyzed (Skin sites) | 57 | 57 | 0
  Post-application 6 | 0 [0 to 0] | 0 [0 to 0] |
  Post-application 7: number analyzed (Participants) | 57 | 57 | 0
  Post-application 7: number analyzed (Skin sites) | 57 | 57 | 0
  Post-application 7 | 0 [0 to 0] | 0 [0 to 0] |
  Post-application 8: number analyzed (Participants) | 57 | 57 | 0
  Post-application 8: number analyzed (Skin sites) | 57 | 57 | 0
  Post-application 8 | 0 [0 to 0] | 0 [0 to 0] |
  Post-application 9: number analyzed (Participants) | 57 | 57 | 0
  Post-application 9: number analyzed (Skin sites) | 57 | 57 | 0
  Post-application 9 | 0 [0 to 0] | 0 [0 to 0] |

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study, ~5 weeks.
Description: Adverse event is presented for all subjects by subject since the event was systemic in nature. Each subject received each treatment (test, positive control, and negative control) at a different skin site over the same study period.
Arm/Group | Test Article (Collagen Wound Dressing) and Negative Control (Distilled Water)
All-Cause Mortality (participants affected / at risk) | 0/86
Serious Adverse Events (participants affected / at risk) | 0/86
Other Adverse Events (participants affected / at risk) | 1/86
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Article (Collagen Wound Dressing) and Negative Control (Distilled Water) (N=86)
headache and stomach pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT06283173/Prot_002.pdf